CLINICAL TRIAL: NCT05760209
Title: SMN Circular RNAs as Potential New Targets and Biomarkers for the Therapeutic Response in Spinal Muscular Atrophy
Brief Title: SMN Circular RNAs as Potential New Targets and Biomarkers for SMA
Acronym: CircSMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4348
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: biomarkers, spinal muscular atrophy; outcome
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spinal Muscular Atrophy (SMA) is a life-threatening disease in infancy that is caused by inactivating mutations in the Survival Motor Neuron 1 (SMN1) gene1,2. SMN1 mutations lead to deficiency in SMN protein, which results in degeneration of motor neurons in the spinal cord, progressive muscle weakness and atrophy. The almost identical SMN2 gene does not suffice SMN function, because skipping of exon 7 in its mRNA yields an unstable protein. Nevertheless, SMN2 represents a disease modifier gene and increasing its expression or rescuing its splicing defect have long been considered elective strategies for SMA1,2. After substantial translational research efforts, the first therapies eliciting clinical benefits for SMA patients have recently become available3. Nusinersen, an antisense oligonucleotide (ASO), and Risdiplasm, a small molecule, bind the SMN2 RNA and promote splicing of exon 7. On the other hand, Zolgesma, an adeno-associated virus delivering the SMN1 gene (scAAV9-SMN), bypasses the need to correct the splicing defect. Nevertheless, none of these therapies currently represents a complete cure for patients, because not all of them respond equally and in a significant portion of patients the symptoms are attenuated but not corrected3. It is believed that early treatment, possibly at a pre-symptomatic stage, would positively affect the clinical response and may significantly improve patient's management. However, another critical point is the current lack of information on the long-term efficacy and safety of the current treatments4. In this scenario, it is likely that further elucidation of the biological functions of the SMN genes and the identification of robust biomarkers for stratification of patients will set the ground for more "personalized" therapies, which may account for the clinical variability observed in patients and help improving the therapies in use.

DETAILED DESCRIPTION:
This project aims at investigating the potential value of SMN circRNAs as biomarkers of SMA, in terms of prediction of disease severity and response to therapeutic treatments.

In particular, we aim to:

1. Evaluate the potential of SMN circRNAs as biomarkers of SMA clinical outcome. We will evaluate which SMN circRNAs are released in body fluids of SMA patients undergoing treatments and whether they display prognostic power as predictors of disease progression and clinical response to therapies.
2. Perform a prospective analysis of SMN circRNAs expression in pre-symptomatic SMA patients. We will analyze the expression levels of SMN circRNAs in body fluids of SMA patients identified by neonatal genetic screening.

The results of our project may identify new tools to better stratify SMA patients and to improve the efficacy of the currently available treatments for this disease.

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of SMA, without any restrictions for phenotype (i.e. presymptomatic patients, SMA 0, SMA I, SMA II, SMA III, SMA IV patients), number of SMN2, age or gender.
* Treatment with Nusinersen or Risdiplam or Zolgensma.

Exclusion Criteria:

unable to provide consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with SMA trewated according to standards of care
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2024-07-21 (Estimated); Study Completion 2024-07-21 (Estimated)

PRIMARY OUTCOMES:
survival motor neuron (SMN) circular RNA | 36 months
  biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Mercuri, Principal Investigator — F Policlinico Gemelli IRCCS
Locations (1):
- Policlinico gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
aggregate data only